CLINICAL TRIAL: NCT03311009
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Ascending Doses of GLPG1972 for 4 Weeks in Subjects With Osteoarthritis
Brief Title: A Study With GLPG1972 in Osteoarthritis Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1972-CL-104
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GLPG1972 (Experimental)
  Interventions: Drug: GLPG1972 cohort 1; Drug: GLPG1972 cohort 2; Drug: GLPG1972 cohort 3
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG1972 cohort 1 — GLPG1972 dose 1 provided as oral tablets q.d.
  Arms: GLPG1972
Drug: GLPG1972 cohort 2 — GLPG1972 dose 2 provided as oral tablets q.d.
  Arms: GLPG1972
Drug: GLPG1972 cohort 3 — GLPG1972 dose 3 provided as oral tablets q.d.
  Arms: GLPG1972
Drug: Placebo — Matching placebo provided as oral tablets q.d.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, stratified, ascending dose, single center study, in three semi-sequential cohorts of 10 male and female subjects of nonchildbearing potential with Osteoarthritis (OA), administered GLPG1972 or placebo. Per cohort, 10 subjects will be randomized in a 4:1 allocation ratio to active treatment with GLPG1972 or matching placebo. In each cohort, OA subjects will be stratified for age (50- 64 years and 65-75 years) with a minimum of 2 of each sex per age group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects of non-childbearing potential, 50-75 years of age on the date of signing the Informed Consent Form (ICF), inclusive extremes.
2. Diagnosis of OA (knee and/or hip) made by their physician based on symptoms, clinical signs and documented historical imaging evidence.
3. A body mass index (BMI) between 18.0 and 34.9 kg/m2, inclusive extremes.
4. Judged to be in age-appropriate good health by the investigator based upon the results of a medical history, physical examination, vital signs and 12-lead ECG, and fasting clinical laboratory profile.
5. Subjects with a stable chronic illness at least 3 months will be accepted subject to the investigator's judgment.

Exclusion Criteria:

1. Administration of intraarticular glucocorticoid injections or hyaluronan injections in the last 3 months prior to study screening.
2. Subjects who underwent or are on a waiting list for total hip or knee replacement and any other surgery planned during the study (up to Day 50).
3. Known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug as determined by the investigator, such as anaphylaxis requiring hospitalization.
4. Positive serology for HBsAg or HCV antibody or history of hepatitis from any cause with the exception of hepatitis A.
5. History of or a current immunosuppressive condition.
6. Clinically significant serious, per investigator's discretion, and/or unstable illness in the 3 months before screening
7. Renal function with an estimated creatinine clearance < 60 mL/min based on the Cockcroft-Gault formula. Retesting is allowed once (see Section 5.2).
8. Use of verapamil, diltiazem, amitriptyline, warfarin, acenocoumarol, phenobarbital and phenytoin, within 4 weeks before first study drug administration
9. Consumption of herbal medications that are strong inhibitors and/or inducers of CYPs (e.g., St. John's Wort) and grapefruit/grapefruit products, Seville oranges, or any poppy seed, within 7 days prior to the first study drug administration.
10. History of solid organ or hematopoietic cell transplantation.
11. History of malignancy within the past 5 years.
12. Clinically significant abnormalities detected on 12-lead ECG of either rhythm or conduction (e.g., QTcF ≥ 450 ms for males and QTcF ≥ 470 ms for females, or a known long QT syndrome).
13. Significant blood loss (including blood donation [> 450 mL]), or transfusion of any blood product within 12 weeks prior to screening

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Difference between GLPG1972 treated subjects and placebo subjects in the number of Adverse Events | From screening until the final follow up visit (day 50)
  To assess safety and tolerability of GLPG1972 in OA patients
Difference in the number of GLPG1972 treated subjects and placebo subjects with abnormal vital signs | From screening until the final follow up visit (day 50)
  To assess safety and tolerability of GLPG1972 in OA patients
Difference in the number of GLPG1972 treated subjects and placebo subjects with abnormal clinical laboratory evaluations | Screening, Days -1, 2, 4, 8, 9, 15, 22, 29, 43 and the final follow up visit (day 50)
  To assess safety and tolerability of GLPG1972 in OA patients
Difference in the number of GLPG1972 treated subjects and placebo subjects with abnormal physical examination | Screening, days -1, 1, 2, 8, 15, 22, 29, 43 and the final follow up visit (day 50
  To assess safety and tolerability of GLPG1972 in OA patients
Difference in the number of GLPG1972 treated subjects and placebo subjects with abnormal ECG | Screening, days 1, 2, 3, 4, 8, 15, 22, 29, 43 and the final follow up visit (day 50)
  To assess safety and tolerability of GLPG1972 in OA patients
Difference in the number of GLPG1972 treated subjects and placebo subjects with abnormal Holter assessment | Day -1 to days 1 and Day 10 to day 11
  To assess safety and tolerability of GLPG1972 in OA patients
The maximum observed plasma concentration of GLPG1972 (Cmax) | Days 1, 2, 3, 4, 6, 8, 10, 15, 16, 22, 29 and 43
  To assess PK of GLPG1972 in OA patients
The time (tmax) to reach Cmax of GLPG1972 | Days 1, 2, 3, 4, 6, 8, 10, 15, 16, 22, 29 and 43
  To assess PK of GLPG1972 in OA patients
The plasma concentration of GLPG1972 24 after the last dose | Days 1, 2, 3, 4, 6, 8, 10, 15, 16, 22, 29 and 43
  To assess PK of GLPG1972 in OA patients
The area under the plasma concentration time curve from time 0 until the last quantifieble dose | Days 1, 2, 3, 4, 6, 8, 10, 15, 16, 22, 29 and 43
  To assess PK of GLPG1972 in OA patients

SECONDARY OUTCOMES:
Percentage reduction of neo-epitope ARGS vs baseline | Days 1, 3, 6, 8, 10, 15, 22, 29, 43 and the final follow up visit (day 50)
  To assess PD of GLPE1972 in OA patients

CONTACTS AND LOCATIONS:
Overall Officials: Ann Fieuw, MD, MSc, Study Director — Galapagos NV
Locations (1):
- Covance Daytona Beach, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen L, Huang FL, Tang Q, Zhao ZK, Ye ZY, Liang JH. Targeted therapy for knee osteoarthritis: From basic to clinics. Medicine (Baltimore). 2025 Aug 15;104(33):e43686. doi: 10.1097/MD.0000000000043686. PMID 40826764